CLINICAL TRIAL: NCT00485836
Title: A Phase III, Multicenter, Randomized, Sham Injection-Controlled Study of the Efficacy and Safety of Ranibizumab Injection Compared With Sham in Subjects With Macular Edema Secondary to Central Retinal Vein Occlusion
Brief Title: A Study of the Efficacy and Safety of Ranibizumab Injection in Patients With Macular Edema Secondary to Central Retinal Vein Occlusion (CRUISE)
Acronym: CRUISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FVF4166g
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: CRVO; RVO; Lucentis; Edema
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion; Edema | interventions — salicylhydroxamic acid; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Sham injection (Sham Comparator)
  Interventions: Drug: Sham injection
- Ranibizumab injection 0.3 mg (Experimental)
  Interventions: Drug: Ranibizumab injection 0.3 mg
- Ranibizumab injection 0.5 mg (Experimental)
  Interventions: Drug: Ranibizumab injection 0.5 mg

INTERVENTIONS:
Drug: Sham injection — Sham injection in a single-dose regimen given every month (Day 0 through the Month 5 visit), for a total of six sham injections.
  Other Names: Lucentis
  Arms: Sham injection
Drug: Ranibizumab injection 0.3 mg — Ranibizumab injection 0.3 mg in a single-dose regimen given every month (Day 0 through the Month 5 visit), for a total of six injections.
  Arms: Ranibizumab injection 0.3 mg
Drug: Ranibizumab injection 0.5 mg — Ranibizumab injection 0.5 mg in a single-dose regimen given every month (Day 0 through the Month 5 visit), for a total of six injections.
  Other Names: Lucentis
  Arms: Ranibizumab injection 0.5 mg

SUMMARY:
This was a Phase III, multicenter, randomized, double-masked, sham injection-controlled study of the efficacy and safety of intravitreal ranibizumab compared with sham injections in patients with macular edema secondary to central retinal vein occlusion (CRVO); 392 patients with CRVO were enrolled at 95 investigational sites in the United States. The study included a treatment period (6 months) and an observation period (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide signed Informed Consent Form
* Age ≥ 18 years
* For sexually active women of childbearing potential, use of an appropriate form of contraception (or abstinence) for the duration of the study
* Ability and willingness to return for all scheduled visits and assessments

Ocular Inclusion Criterion (Study Eye):

* Foveal center-involved macular edema secondary to CRVO
* BCVA using ETDRS charts of 20/40 to 20/320 (Snellen equivalent)
* Mean central subfield thickness ≥ 250 μm on two optical coherence tomography (OCT) measurements (at screening [confirmed by the central reading center] and Day 0 [confirmed by the evaluating physician])
* Media clarity, pupillary dilation, and participant cooperation sufficient to obtain adequate fundus photographs

Exclusion Criteria:

* History of cerebral vascular accident or myocardial infarction within 3 months prior to Day 0
* History of any anti-vascular endothelial growth factor (VEGF) or treatment in the fellow eye within 3 months prior to Day 0
* History of any systemic anti-VEGF or pro-VEGF treatment within 6 months prior to Day 0
* History of allergy to fluorescein
* History of allergy to ranibizumab injection or related molecule
* Relevant systemic disease that may be associated with increased systemic VEGF levels (namely, all active malignancies); history of successfully treated malignancies is not an exclusion criterion.
* Uncontrolled blood pressure
* Pregnancy or lactation
* Any condition that, in the opinion of the investigator, would preclude participation in the study (e.g., chronic alcoholism or drug abuse, personality disorder or use of major tranquilizers, indicated difficulty in long-term follow-up, and likelihood of survival of less than 1 year)
* Participation in an investigational trial within 30 days prior to Day 0 that involved treatment with any drug (excluding vitamins and minerals) or device that has not received regulatory approval at time of study entry

Ocular Exclusion Criteria (Study Eye):

* Prior episode of retinal vein occlusion (RVO)
* Brisk afferent pupillary defect
* History of radial optic neurotomy or sheathotomy
* History or presence of age-related macular degeneration (AMD; dry or wet form)
* History of any anti-VEGF treatment in the study eye within 3 months prior to Day 0
* History of laser photocoagulation for macular edema within 4 months prior to Day 0
* History of panretinal scatter photocoagulation or sector laser photocoagulation within 3 months prior to randomization or anticipated within the next 4 months following randomization
* History of intraocular corticosteroid use within 3 months prior to Day 0
* History of pars plana vitrectomy
* History of intraocular surgery (including cataract extraction, scleral buckle, etc.) within 2 months prior to Day 0 or anticipated within the next 7 months following Day 0
* History of yttrium-aluminum-garnet capsulotomy performed within 2 months prior to Day 0
* Previous filtration surgery in the study eye
* History of herpetic ocular infection
* History of ocular toxoplasmosis
* History of rhegmatogenous retinal detachment
* History of idiopathic central serous chorioretinopathy
* Evidence upon examination of vitreoretinal interface disease (e.g., vitreomacular traction, epiretinal membrane), either on clinical examination or OCT, thought to be contributing to macular edema
* An eye that, in the investigator's opinion, would not benefit from resolution of macular edema, such as eyes with foveal atrophy, dense pigmentary changes, or dense subfoveal hard exudates
* Presence of an ocular condition that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the study (e.g., uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass syndrome, or prior macula-off rhegmatogenous retinal detachment)
* Visually significant hemorrhage obscuring the fovea and felt to be a major contributor to reduced visual acuity
* Presence of a substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., a 20/40 cataract)
* Aphakia
* Relevant ocular disease that may be associated with increased intraocular VEGF levels (namely, uveitis, neovascular glaucoma, neovascular AMD, diabetic retinopathy, diabetic maculopathy, or ocular ischemic syndrome)
* Improvement of > 10 letters on best corrected visual acuity (BCVA) between screening and Day 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Rubio, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Suner IJ, Bressler NM, Varma R, Lee P, Dolan CM, Ward J, Colman S, Rubio RG. Reading speed improvements in retinal vein occlusion after ranibizumab treatment. JAMA Ophthalmol. 2013 Jul;131(7):851-6. doi: 10.1001/jamaophthalmol.2013.114. PMID 23699977
- [Derived] Bhisitkul RB, Campochiaro PA, Shapiro H, Rubio RG. Predictive value in retinal vein occlusions of early versus late or incomplete ranibizumab response defined by optical coherence tomography. Ophthalmology. 2013 May;120(5):1057-63. doi: 10.1016/j.ophtha.2012.11.011. Epub 2013 Feb 14. PMID 23415775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Please note that although the table below is titled "Overall Study," the completion rates are for the 6-month Treatment Period only (i.e., does not include the 6-month Observation Period data).
Period: Overall Study
Arm/Group | Sham Injection | Ranibizumab Injection 0.3 mg | Ranibizumab Injection 0.5 mg
Started | 130 | 132 | 130
Received Study Drug (Safety Population) | 129 | 132 | 129
Completed | 115 | 129 | 119
Not Completed | 15 | 3 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Injection | Ranibizumab Injection 0.3 mg | Ranibizumab Injection 0.5 mg | Total
Number analyzed (Participants) | 130 | 132 | 130 | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (13.1) | 69.7 (11.6) | 67.6 (12.4) | 67.6 (12.5)
Age, Customized [Number; unit: participants]
  < 45 years | 10 | 5 | 5 | 20
  45 to < 65 years | 50 | 36 | 46 | 132
  65 to < 85 years | 67 | 80 | 71 | 218
  ≥ 85 years | 3 | 11 | 8 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 61 | 50 | 169
  Male | 72 | 71 | 80 | 223

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Score at 6 Months
Description: BCVA score in the study eye was based on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity charts (number of correct letters) and assessed at a starting distance of 4 meters.
Time Frame: Baseline and 6 months
Population: Intent to treat (randomized) population. Missing values were imputed using the last-observation-carried-forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sham Injection | Ranibizumab Injection 0.3 mg | Ranibizumab Injection 0.5 mg
Number analyzed (Participants) | 130 | 132 | 130
Units on a scale
  Baseline | 49.2 (14.7) | 47.4 (14.8) | 48.1 (14.6)
  Mean Change from Baseline at Month 6 | 0.8 (16.2) | 12.7 (15.9) | 14.9 (13.2)
Statistical Analysis 1: Comparison: Sham Injection vs Ranibizumab Injection 0.3 mg; Test type: Superiority or Other; p < 0.0001, ANOVA — The Hochberg-Bonferroni multiple comparison procedure was used to adjust for comparisons of the two ranibizumab groups with the sham-injection group to maintain an overall type I error rate of 0.05; Stratified by baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters); Difference in Least Squares means = 11.5, 95% CI [7.7 to 15.3]
Statistical Analysis 2: Comparison: Sham Injection vs Ranibizumab Injection 0.5 mg; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Stratified by baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters); Difference in Least Squares means = 13.8, 95% CI [10.3 to 17.4]

2. Secondary Outcome: Percentage of Participants Who Gained ≥ 15 Letters in BCVA Score at Month 6 Compared With Baseline
Description: BCVA score based on the ETDRS visual acuity charts (number of correct letters) and assessed at a starting distance of 4 meters.
Time Frame: Baseline and 6 months
Population: Intent to treat (randomized) population. Missing values were imputed using the LOCF method.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sham Injection | Ranibizumab Injection 0.3 mg | Ranibizumab Injection 0.5 mg
Number analyzed (Participants) | 130 | 132 | 130
Percentage of participants | 16.9 [10.5 to 23.4] | 46.2 [37.7 to 54.7] | 47.7 [39.1 to 56.3]
Statistical Analysis 1: Comparison: Sham Injection vs Ranibizumab Injection 0.3 mg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel χ²; Stratified by baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters); Difference in percentage = 29.3, 95% CI [18.8 to 39.7] — Weighted estimates adjusted for baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters) using Cochran-Mantel-Haenszel weights
Statistical Analysis 2: Comparison: Sham Injection vs Ranibizumab Injection 0.5 mg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel χ²; Stratified by baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters); Difference in percentage = 30.3, 95% CI [19.6 to 40.9] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants Who Lost < 15 Letters in BCVA Score at Month 6 Compared With Baseline
Description: as for outcome 2
Time Frame: Baseline and 6 months
Population: Intent to treat (randomized) population. Missing values were imputed using the LOCF method.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sham Injection | Ranibizumab Injection 0.3 mg | Ranibizumab Injection 0.5 mg
Number analyzed (Participants) | 130 | 132 | 130
Percentage of participants | 84.6 [78.4 to 90.8] | 96.2 [93.0 to 99.5] | 98.5 [96.3 to 100]
Statistical Analysis 1: Comparison: Sham Injection vs Ranibizumab Injection 0.3 mg; Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel χ²; Stratified by baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters); Difference in percentage = 11.3, 95% CI [4.3 to 18.2] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Sham Injection vs Ranibizumab Injection 0.5 mg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel χ²; Stratified by baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters); Difference in percentage = 13.6, 95% CI [7.2 to 20.1] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants With a Central Foveal Thickness of ≤ 250 μm at Month 6
Description: A central reading center assessed all optical coherence tomography (OCT) images. Central foveal thickness was defined as the center point thickness.
Time Frame: 6 months
Population: Intent to treat (randomized) population. Missing values were imputed using the LOCF method.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sham Injection | Ranibizumab Injection 0.3 mg | Ranibizumab Injection 0.5 mg
Number analyzed (Participants) | 130 | 132 | 130
Percentage of participants | 23.1 [15.8 to 30.3] | 75.0 [67.6 to 82.4] | 76.9 [69.7 to 84.2]
Statistical Analysis 1: Comparison: Sham Injection vs Ranibizumab Injection 0.3 mg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel χ²; Stratified by baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters); Difference in percentage = 51.9, 95% CI [41.6 to 62.3] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Sham Injection vs Ranibizumab Injection 0.5 mg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel χ²; Stratified by baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters); Difference in percentage = 54.0, 95% CI [44.0 to 64.1] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Mean Absolute Change From Baseline in Central Foveal Thickness at Month 6
Description: A central reading center assessed all OCT images. Central foveal thickness was defined as the center point thickness.
Time Frame: Baseline and 6 months
Population: Intent to treat (randomized) population. Missing values were imputed using the LOCF method.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Sham Injection | Ranibizumab Injection 0.3 mg | Ranibizumab Injection 0.5 mg
Number analyzed (Participants) | 129 | 131 | 130
μm
  Baseline | 687.0 (237.6) | 679.9 (242.2) | 688.7 (253.1)
  Mean Absolute Change from Baseline at Month 6 | -167.7 (308.4) | -433.7 (295.9) | -452.3 (257.6)
Statistical Analysis 1: Comparison: Sham Injection vs Ranibizumab Injection 0.3 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Pairwise ANCOVA models adjusted for baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters) and baseline value of central foveal thickness; Difference in Least Squares means = -272.2, 95% CI [-329.9 to -214.5]
Statistical Analysis 2: Comparison: Sham Injection vs Ranibizumab Injection 0.5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 5, analysis 1]; Difference in Least Squares means = -283.8, 95% CI [-337.8 to -229.8]

6. Secondary Outcome: Mean Change From Baseline in the National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25) Near Activities Subscale Score at Month 6
Description: The NEI VFQ-25 (v. 2000; Interviewer Format) consisted of the base set of 25 questions, plus the optional additional questions (where questions A3, A4, and A5 pertained to the Near Activities Subscale). Scores ranged from 0 to 100; a higher score represented better functioning.
Time Frame: Baseline and 6 months
Population: Intent to treat (randomized) population; however, patients without a baseline score were excluded from analysis.
Measure: Mean (Standard Deviation); unit: Points on the NEI VFQ-25 subscale
Arm/Group | Sham Injection | Ranibizumab Injection 0.3 mg | Ranibizumab Injection 0.5 mg
Number analyzed (Participants) | 127 | 130 | 128
Points on the NEI VFQ-25 subscale
  Baseline at Month 6 | 69.9 (22.6) | 71.2 (22.2) | 70.7 (20.3)
  Change from baseline at Month 6 | 5.1 (17.1) | 10.2 (17.4) | 9.3 (18.1)
Statistical Analysis 1: Comparison: Sham Injection vs Ranibizumab Injection 0.3 mg; Test type: Superiority or Other; p = 0.0019, ANCOVA; Pairwise ANCOVA models adjusted for baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters) and baseline Near Activities Subscale score; Difference in Least Squares means = 5.8, 95% CI [2.1 to 9.4]
Statistical Analysis 2: Comparison: Sham Injection vs Ranibizumab Injection 0.5 mg; Test type: Superiority or Other; p = 0.0099, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference in Least Squares means = 4.9, 95% CI [1.2 to 8.6]

7. Secondary Outcome: Mean Change From Baseline in the NEI VFQ-25 Distance Activities Subscale Score at Month 6
Description: The NEI VFQ-25 (v. 2000; Interviewer Format) consisted of the base set of 25 questions, plus the optional additional questions (where questions A6, A7, and A8 pertained to the Distance Activities Subscale). Scores ranged from 0 to 100; a higher score represented better functioning.
Time Frame: Baseline and 6 months
Population: Intent to treat (randomized) population; however, patients without a baseline score were excluded from analysis.
Measure: Mean (Standard Deviation); unit: Points on the NEI VFQ-25 subscale
Arm/Group | Sham Injection | Ranibizumab Injection 0.3 mg | Ranibizumab Injection 0.5 mg
Number analyzed (Participants) | 127 | 130 | 128
Points on the NEI VFQ-25 subscale
  Baseline at Month 6 | 77.0 (22.5) | 77.3 (19.8) | 77.0 (19.7)
  Change from baseline at Month 6 | 2.8 (15.6) | 8.9 (13.7) | 6.7 (16.3)
Statistical Analysis 1: Comparison: Sham Injection vs Ranibizumab Injection 0.3 mg; Test type: Superiority or Other; p = 0.0002, ANCOVA; Pairwise ANCOVA models adjusted for baseline visual acuity score (≤ 34, 35-54, ≥ 55 letters) and baseline Distance Activities Subscale score; Difference in Least Squares means = 6.3, 95% CI [3.1 to 9.5]
Statistical Analysis 2: Comparison: Sham Injection vs Ranibizumab Injection 0.5 mg; Test type: Superiority or Other; p = 0.0199, ANCOVA; [statistical method as in outcome 7, analysis 1]; Difference in Least Squares means = 4.1, 95% CI [0.7 to 7.6]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Investigators assessed the occurrence of AE/SAEs at all study visits. Summaries are for the safety-evaluable population and include events regardless of relation to study drug or location (e.g. non-study eye events are included). For each AE/SAE, the number of patients experiencing the event, not the number of occurrences of the event, is reported.
Arm/Group | Sham Injection | Ranibizumab Injection 0.3 mg | Ranibizumab Injection 0.5 mg
Serious Adverse Events (participants affected / at risk) | 13/129 | 16/132 | 13/129
Other Adverse Events (participants affected / at risk) | 116/129 | 113/132 | 111/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection (N=129) | Ranibizumab Injection 0.3 mg (N=132) | Ranibizumab Injection 0.5 mg (N=129)
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 2 | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 1 | 0
Blindness Unilateral (Eye disorders) | 0 | 0 | 1
Vitreous Hemorrhage (Eye disorders) | 1 | 0 | 0
Corneal Edema (Eye disorders) | 0 | 1 | 0
Iris Neovascularization (Eye disorders) | 0 | 0 | 1
Retinal Disorder (Eye disorders) | 0 | 1 | 0
Macular Ischemia (Eye disorders) | 1 | 0 | 0
Retinal Artery Occlusion (Eye disorders) | 0 | 1 | 0
Retinal Vascular Disorder (Eye disorders) | 0 | 1 | 0
Retinal Vascular Occlusion (Eye disorders) | 0 | 0 | 1
Retinal Vein Occlusion (Eye disorders) | 2 | 1 | 1
Maculopathy (Eye disorders) | 0 | 1 | 0
Retinal Depigmentation (Eye disorders) | 0 | 1 | 0
Macular Edema (Eye disorders) | 2 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 1 | 0
Food Allergy (Immune system disorders) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Lead Dislodgement (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 2 | 0
Transient Ischemic Attack (Nervous system disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 0
Venous Occlusion (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection (N=129) | Ranibizumab Injection 0.3 mg (N=132) | Ranibizumab Injection 0.5 mg (N=129)
Conjunctival Hemorrhage (Eye disorders) | 43 | 57 | 53
Eye Irritation (Eye disorders) | 6 | 6 | 10
Eye Pain (Eye disorders) | 14 | 12 | 24
Foreign Body Sensation in Eyes (Eye disorders) | 5 | 4 | 9
Iris Neovascularization (Eye disorders) | 9 | 2 | 1
Macular Edema (Eye disorders) | 11 | 7 | 4
Maculopathy (Eye disorders) | 13 | 21 | 19
Myodesopsia (Eye disorders) | 5 | 9 | 12
Ocular Vascular Disorder (Eye disorders) | 0 | 2 | 8
Optic Disc Vascular Disorder (Eye disorders) | 8 | 7 | 2
Retinal Depigmentation (Eye disorders) | 8 | 12 | 10
Retinal Exudates (Eye disorders) | 18 | 36 | 25
Retinal Hemorrhage (Eye disorders) | 17 | 15 | 16
Retinal Pigmentation (Eye disorders) | 4 | 7 | 2
Retinal Vascular Disorder (Eye disorders) | 19 | 21 | 19
Vitreous Detachment (Eye disorders) | 6 | 1 | 8
Vitreous Hemorrhage (Eye disorders) | 8 | 5 | 7
Nasopharyngitis (Infections and infestations) | 3 | 8 | 7
Intraocular Pressure Increased (Investigations) | 5 | 11 | 11
Hypertension (Vascular disorders) | 8 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.